CLINICAL TRIAL: NCT01308983
Title: Study of Amiloride on Vascular Phenotypes in Young Adults With Prehypertension
Acronym: SAPHA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Yanbin Dong, Professor, Department of Pediatrics, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1000
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Prehypertension
Keywords: Prehypertension; Flow mediated dilation; Pulse wave velocity; carotid compliance; Prehypertension and amiloride
MeSH Terms: conditions — Prehypertension | interventions — Amiloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Amiloride (Other)
  Interventions: Drug: Amiloride

INTERVENTIONS:
Drug: Amiloride — Amiloride 10 mg orally once a day for 16 weeks

SUMMARY:
Primary Specific Aim: To test the hypothesis that amiloride will improve vascular health of young adults with prehypertension.

ELIGIBILITY:
Inclusion Criteria:

* Prehypertensive: Having systolic BP between 120 to 139 mmHg and/or diastolic BP between 80 to 89 mmHg during screening visit. BP will be measured manually tree times at 10 minutes interval after subjects sit quietly for at least 5 minutes in a chair. The average of last two BP measurements will be taken into consideration.
* Male or female of Caucasian or African-American origin.
* No history of any major past and current medical illness (such as diabetes, renal disease, liver disease etc.)
* Not taking any medication that affects blood pressure.

Exclusion Criteria:

* HbA1C > 7.0 % during screening visit.
* Serum potassium > 5.5 mEq/L during screening and/or any testing visit due to risk of developing hyperkalemia.
* Serum creatinine > 1.5 mg/100 ml and/or creatinine clearance < 50 ml/min* (Glomerular Filtration Rate Estimate by Abbreviated MDRD Study Equation)35 during screening and/or any testing visit due to risk of developing renal dysfunction.
* Female having positive pregnancy test during screening and/or any testing visit.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Vascular phenotypes | 16 weeks
  (Flow mediated dilation, Pulse wave velocity, and carotid artery compliance)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgia Prevention Institute, Augusta, Georgia, United States

REFERENCES:
- [Derived] Bhagatwala J, Harris RA, Parikh SJ, Zhu H, Huang Y, Kotak I, Seigler N, Pierce GL, Egan BM, Dong Y. Epithelial sodium channel inhibition by amiloride on blood pressure and cardiovascular disease risk in young prehypertensives. J Clin Hypertens (Greenwich). 2014 Jan;16(1):47-53. doi: 10.1111/jch.12218. Epub 2013 Oct 31. PMID 24410943